CLINICAL TRIAL: NCT06328582
Title: Clinical Effect of Acupuncture Technique for Restoring Consciousness Combined With Scalp Acupuncture on Post-stroke Dysphagia
Brief Title: Acupuncture Technique for Restoring Consciousness on Post-stroke Dysphagia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, The Research Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Zhenjiu Post-stroke dysphagia
Record Dates: First submitted 2024-03-08; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine treatment+Acupuncture Technique for Restoring Consciousness Combined with Scalp Acupuncture (Experimental): The experimental group was given routine treatment. Moreover, the experimental group will receive Acupuncture Technique for Restoring Consciousness.
  Interventions: Behavioral: Routine rehabilitation training; Procedure: Acupuncture Technique for Restoring Consciousness combined with Scalp Acupuncture
- routine treatment (Active Comparator): The experimental group was given routine treatment.
  Interventions: Behavioral: Routine rehabilitation training

INTERVENTIONS:
Behavioral: Routine rehabilitation training — Balance function training: Patients were instructed to achieve weight shift between the left and right sides of the balance bar in a standing position.
  Walking function training: based on hip, knee, and ankle control training, patients were instructed to take steps training.
  Core muscle strength training: Patients were instructed to maintain 3 minutes of training in Bridge-style movement.
  Functional training of daily living: including training on dressing and undressing, independent eating, painting, and writing.
Procedure: Acupuncture Technique for Restoring Consciousness combined with Scalp Acupuncture — Acupuncture Technique for Restoring Consciousness:
  Main acupoints: Neiguan (bilateral), Renzhong, Sanyinjiao (affected side) Additional acupoints: Fengchi, Wangu, Yifeng (bilateral), and posterior pharyngeal wall needling.
  Scalp Acupuncture Method:
  Based on the standard treatment lines for scalp acupuncture [17], select the anterior oblique line of vertex-temporal region, posterior oblique line of vertex-temporal region, and anterior line of temporal region (bilateral).
  Arms: routine treatment+Acupuncture Technique for Restoring Consciousness Combined with Scalp Acupuncture

SUMMARY:
This is a randomized controlled study, including post-stroke dysphagic patients. The participants were divided randomly into the experimental group and the control group. Both two groups were given routine treatment and swallowing rehabilitation training. Moreover, the experimental group was given Acupuncture Technique for Restoring Consciousness. Swallowing function will be compared before and after treatment.

DETAILED DESCRIPTION:
This is a randomized controlled study, including post-stroke dysphagic patients. The participants were divided randomly into the experimental group and the control group. Both two groups were given routine treatment and swallowing rehabilitation training. Moreover, the experimental group was given Acupuncture Technique for Restoring Consciousness. Swallowing function will be compared before and after treatment.

Specifically, our main focus is on Neiguan, Renzhong and Sanyinjiao.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Meeting the diagnostic criteria for stroke.
* Diagnosed with dysphagia confirmed by the video fluoroscopic swallowing study.
* Water swallow test> Level 3.
* Stable vital signs, conscious, able to cooperate with assessment and treatment.

Exclusion Criteria:

* Dysphagia possibly caused by other reasons, such as cerebrovascular disease, trauma, neuromuscular diseases, malignant diseases of the pharynx and larynx, and digestive tract diseases.
* History of mental diseases or use of antipsychotics.
* Complicated with cognitive impairment or consciousness dysfunction.
* Simultaneously suffering from severe liver, kidney failure, tumors, or hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | day 1 and day 28
  The Penetration-Aspiration Scale was conducted under video fluoroscopic swallowing study. The scale is a standardized tool used to assess the safety of swallowing. The scale was developed to evaluate the entry of material into the airway (penetration) and the subsequent passage of material below the vocal folds (aspiration) during swallowing. The scale ranges from 1 to 8, with each level representing different degrees of penetration or aspiration.

SECONDARY OUTCOMES:
Functional Oral Intake Scale | day 1 and day 28
  The scale reflects the patient's oral intake. Studies have shown that this scale can also serve as an independent measure of intake for post-stroke dysphagia patients. The scale is divided into 7 levels, with the level positively correlated with swallowing function. Level 7 indicates normal swallowing function.
Gugging Swallowing Screen | day 1 and day 28
  Gugging Swallowing Screen is a safe and simple bedside screening tool that consists of 2 testing parts. It can accurately assess the risk of aspiration and differentiate between different food consistencies. The scale can not only detect the risk of aspiration in patients but also guide their diet. The scale has a maximum score of 20, indicating normal swallowing function. The lower the score, the more severe the swallowing disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Chair — Site Coordinator of United Medical Group